CLINICAL TRIAL: NCT07112807
Title: Comparison of the Effects of ShoulderSphere Exercises and Bodyblade Exercises in Young Individuals With Asymptomatic Scapular Dyskinesis: A Randomized Controlled Study
Brief Title: Comparison of the Effects of ShoulderSphere Exercises and Bodyblade Exercises
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Tuğçe Çoban, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-77082166-604.01-975466
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Scapular Dyskinesis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Experimental): Individuals assigned to the control group will be administered resistive exercises targeting the middle and lower trapezius and serratus anterior muscles. The program will progress by increasing the number of exercises and the amount of resistance.
  Interventions: Other: Strengthening Exercises
- ShoulderSphere (Experimental): In addition to the exercises in the control group, exercises will be performed using the ShoulderSphere in the frontal, sagittal and transverse planes.
  Interventions: Other: Strengthening Exercises; Other: ShoulderSphere Exercises and Resistive Exercises
- Bodyblade (Experimental): In addition to the exercises performed in the control group, 15 minutes of exercises using the Bodyblade will be performed. Individuals will perform oscillation exercises in the frontal, sagittal, and transverse planes.
  Interventions: Other: Strengthening Exercises; Other: Bodyblade Exercises and Resistive Exercises

INTERVENTIONS:
Other: Strengthening Exercises — Strengthening exercises targeting the middle and lower trapezius and serratus anterior muscles will be performed. The program will progress by increasing the number of exercises and the amount of resistance.
Other: ShoulderSphere Exercises and Resistive Exercises — In addition to strengthening exercises, exercises will be performed using the ShoulderSphere in the frontal, sagittal and transverse planes with the shoulders in 90° flexion and the elbows in extension.
  Arms: ShoulderSphere
Other: Bodyblade Exercises and Resistive Exercises — In addition to strengthening exercises, 15 minutes of exercises using the Bodyblade will be performed. Individuals will perform oscillation exercises in the frontal, sagittal, and transverse planes while holding the Bodyblade bar firmly with their shoulders in 90° flexion and elbows in extension.
  Arms: Bodyblade

SUMMARY:
The scapula functions as a bridge connecting the upper extremity and the trunk. It contributes to more efficient and functional upper extremity movements. Scapular dyskinesis, defined as a deviation from the resting position and movements of the scapula, can reduce shoulder proprioception, scapular muscle endurance, and upper extremity function. The aim is to compare the long-term effects of exercises performed using the ShoulderSphere and the Bodyblade, which provide oscillatory stimulation and vibration, enhancing neuromuscular control that improves these factors. Forty-five volunteers with asymptomatic scapular dyskinesis will be randomized into three groups. The control group will receive resistive scapular muscle exercises. The ShoulderSphere group will receive exercises performed using the ShoulderSphere in addition to the control group. The Bodyblade group will receive exercises performed using the Bodyblade in addition to the control group. Pre- and post-treatment proprioception, muscle endurance, and upper extremity function will be assessed, and the groups will be compared. The study results will analyze which method is more effective in the rehabilitation program of individuals with asymptomatic scapular dyskinesis and determine its inclusion in the rehabilitation program.

DETAILED DESCRIPTION:
The scapula functions as a critical biomechanical and neuromuscular bridge between the upper extremity and the trunk, playing a key role in shoulder stability and movement efficiency. Proper scapular motion and positioning are essential for optimal upper limb function. Scapular dyskinesis, defined as an alteration in the resting position or dynamic movement of the scapula, is associated with impaired proprioception, decreased endurance of scapular stabilizer muscles, and reduced functional capacity of the upper extremity. Even in asymptomatic individuals, scapular dyskinesis may predispose to future shoulder pathologies if left unaddressed.

In recent years, rehabilitation strategies have increasingly focused on enhancing neuromuscular control and sensorimotor integration through tools that provide oscillatory and vibratory stimuli. Two such tools-ShoulderSphere and Bodyblade-have gained attention for their ability to activate deep stabilizing musculature and improve dynamic scapular control. These devices generate multidirectional resistance and stimulate rapid afferent feedback mechanisms, promoting more efficient and coordinated muscle responses.

In this study, investigating the long-term effects of ShoulderSphere and Bodyblade training in individuals with asymptomatic scapular dyskinesis may provide valuable insight into their therapeutic potential. The study will involve 45 volunteers who will be randomly assigned to three groups. The control group will perform traditional resistive exercises targeting scapular stabilizers. The ShoulderSphere group will receive the same exercise program with the addition of ShoulderSphere-based training. Similarly, the Bodyblade group will perform the standard exercises along with Bodyblade training. Through this comparison, the study aims to determine which intervention offers greater benefits in improving scapular control, proprioception, and upper extremity function over time.

ELIGIBILITY:
Inclusion Criteria:

* Having scapular dyskinesia
* No shoulder or neck pain

Exclusion Criteria:

* Positive Neer, Jobe, or Hawkins tests
* Shoulder instability
* Painful arch during arm elevation
* Painful passive or resisted shoulder external rotation at 90° shoulder abduction
* History of shoulder fracture or surgery
* Presence of shoulder pain in the last 6 months
* Presence of cognitive or neurological impairment

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-08-29 (Estimated); Study Completion 2025-09-12 (Estimated)

PRIMARY OUTCOMES:
Proprioception | Before and after 4 weeks intervention
  Shoulder joint proprioception will be assessed with a digital inclinometer in flexion, abduction, and external rotation.
Scapular Muscle Endurance | Before and after 4 weeks intervention
  Serratus anterior and trapezius muscle endurance will be assessed using a dynamometer.
Upper Extremity Function | Before and after 4 weeks intervention
  The Closed Kinetic Chain Upper Extremity Stability test will be used.
Lateral scapular slide test | Before treatment
  This test will be evaluated to detect scapular dyskinesis.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğçe Çoban, MSc, Study Director — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kibler WB, Sciascia A. Current concepts: scapular dyskinesis. Br J Sports Med. 2010 Apr;44(5):300-5. doi: 10.1136/bjsm.2009.058834. Epub 2009 Dec 8. PMID 19996329
- [Background] Cho J, Lee K, Kim M, Hahn J, Lee W. The Effects of Double Oscillation Exercise Combined with Elastic Band Exercise on Scapular Stabilizing Muscle Strength and Thickness in Healthy Young Individuals: A Randomized Controlled Pilot Trial. J Sports Sci Med. 2018 Mar 1;17(1):7-16. eCollection 2018 Mar. PMID 29535573
- [Background] Lister JL, Del Rossi G, Ma F, Stoutenberg M, Adams JB, Tobkin S, Signorile JF. Scapular stabilizer activity during Bodyblade, cuff weights, and Thera-Band use. J Sport Rehabil. 2007 Feb;16(1):50-67. doi: 10.1123/jsr.16.1.50. PMID 17699887
- [Background] Savitzky JA, Abrams LR, Galluzzo NA, Ostrow SP, Protosow TJ, Liu SA, Handrakis JP, Friel K. Effects of a Novel Rotator Cuff Rehabilitation Device on Shoulder Strength and Function. J Strength Cond Res. 2021 Dec 1;35(12):3355-3363. doi: 10.1519/JSC.0000000000003347. PMID 35133996